CLINICAL TRIAL: NCT06010693
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase 3 Clinical Study to Investigate the Efficacy and Safety of 50 mg Daridorexant in Adult and Elderly Chinese Patients With Insomnia Disorder.
Brief Title: A Study of Daridorexant in Chinese Patients With Insomnia Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0808-301
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2023-08

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daridorexant (Experimental): Participants will receive one daridorexant 50 mg tablet,orally, once daily for about 28 consecutive night on each night approximately 30 minutes before participants intends to try to sleep.
  Interventions: Drug: Daridorexant
- Placebo (Placebo Comparator): Participants will receive one placebo matched to daridorexant 50 mg tablet,orally, once daily for about 28 consecutive night on each night approximately 30 minutes before participants intends to try to sleep.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant — Participants will receive one Daridorexant 50mg tablet, orally, once daily for about 28 consecutive night on each night approximately 30mintues before participants intends to try to sleep.
  Arms: Daridorexant
Drug: Placebo — Participants will receive one placebo matched to daridorexant 50 mg tablet , orally, once daily for about 28 consecutive nights on each night approximately 30mintues before participants intends to try to sleep.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of 50 mg daridorexant in adult and elderly chinese patients with insomnia disorder.

Efficacy will be evaluated on objective and subjective sleep parameters .

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female aged ≥ 18 years old, ≤75 years old.
3. Insomnia disorder according to diagnostic and statistical Manual of Mental Disorder, Fifth Edition (DSM-5®) criteria, as follows:

   3.1 The predominant complaint is dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms:
   * Difficulty initiating sleep
   * Difficulty maintaining sleep, characterized by frequent awakenings or problems returning to sleep after awakenings.
   * Early-morning awakening with inability to return to sleep. 3.2 The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning.

   3.3 The sleep difficulty occurs despite adequate opportunity for sleep. 3.4 The insomnia is not better explained by another sleep-wake disorder (e.g., narcolepsy, a breathing-related sleep disorder, a circadian rhythm sleep-wake disorder, a parasomnia).

   3.5 The insomnia is not attributable to the physiological effects of a substance (e. g., a drug of abuse, a medication) 3.6 Coexisting mental disorders and medical conditions do not adequately explain the predominant complaint of insomnia.

   3.7 Self-reported history of all the following on at least 3 nights per week and for at least 3 months prior to Visit 1: 3.7.1 ≥30 min to fall asleep, and 3.7.2 Wake time during sleep ≥ 30 min, and 3.7.3 Subjective Total Sleep Time (sTST)≤6.5 h
4. Insomnia Severity Index© score≥15
5. Ability to communicate well with the investigator, to understand the study requirements and independently complete the study, as judged by the investigator, to be alert and oriented to person, place, time, and situation.
6. Meeting all the following sleep parameters on at least 3 nights out of 7 nights on the eDiary completed at home between Visit 3 and Visit 4:

   6.1 ≥ 30 min to fall asleep, and 6.2 Wake time during sleep ≥ 30 min, and 6.3 sTST of ≤ 6.5 h
7. Usual bedtime between 20:30 and 00:30 as reported on sleep diary completed between Visit 3 and Visit 4.
8. Regular time in bed between 6 and 9 h as reported on sleep diary completed between Visit 3 and Visit 4.
9. Meeting all the following sleep parameters on the 2 PSG nights at Visit 4:

   9.1 Mean Latency to Persistent Sleep (LPS) ≥ 20 min (with neither of the two nights < 15 min), and 9.2 Mean Wake After Sleep Onset (WASO) ≥ 30 min (with neither of the two nights < 20 min), and 9.3 Mean Total Sleep Time (TST) < 420 min
10. For women of childbearing potential, the following are required:

    * Negative serum pregnancy test (Visit 1).
    * Negative urine pregnancy test (Visit 3, Visit 5).
11. Female and male subjects agree to use the contraception scheme as required by the protocol from Screening visit up to at least 30 days after last D B study treatment intake, and have no plans to become pregnant, planned parenthood or sperm/egg donation plans, unless they have been sterilization surgically (with surgery at least 1 month before dosing), or female are postmenopausal (female subjects with natural menopause ≥12 months, ≥ 50 years old, can be considered postmenopausal after exclusion of pregnancy and other disorders that may cause amenorrhea; If age <50 years by follicle stimulating hormone level confirmed).

Exclusion Criteria:

1. Chronic obstructive pulmonary disease, or any lifetime history of sleep-related breathing disorderlike sleep apnea.
2. Cognitive behavioral therapy (CBT) for any indication is allowed only if the CBT started at least 1 month prior to Visit 4 and the subject agrees to continue this CBT throughout the study.
3. Self-reported usual daytime napping ≥ 1 h per day, and ≥ 3 days per week.
4. Acute or unstable psychiatric conditions (including but not restricted to anxiety disorder, major depression, bipolar disorder, schizophrenia, obsessive compulsive disorder, or depression) that are diagnosed by the Mini International Neuropsychiatric Interview© or that require pharmacological treatment for these disorders. N.B.: subjects with a history of major depressive disorder currently without any symptoms and not requiring treatment are eligible.
5. Mini Mental State Examination© score < 25 in subjects ≥ 50 years.
6. Shift work within 2 weeks prior to the screening visit, or planned shift work during the study.
7. Travel across ≥ 3 time zones within 2 weeks prior to the screening visit, or planned travel across ≥ 3 time zones during the study.
8. Treatment with central nervous system-active drugs, including over-the- counter medication and herbal medicines, are prohibited by this protocol within 5 half-lives of the respective drug (or 2 weeks, whichever is longer) prior to Visit 1, and until 24 h after the end of treatment (the end of the run-out period).
9. Diagnosis of alcohol or substance use disorder within 2 years prior to the screening visit or inability to refrain from drinking alcohol for at least 3 consecutive days.
10. Heavy tobacco use (at least one pack of cigarettes a day or inability to refrain from smoking during the night).
11. Caffeine consumption ≥ 600 mg per day or any caffeine consumption after 4 pm
12. Use of traditional Chinese medicine as prophylaxis or treatment of sleep disturbance within 4 weeks prior to Visit 1 and during the treatment phase.
13. Treatment with another investigational drug within 3 months prior to Visit 1, previous treatment with daridorexant or other orexin receptor antagonists (i.e. lemborexant, YZJ-1139) or previous randomization in any trial involving daridorexant
14. Known hypersensitivity or contraindication to drugs of the same class as the study treatment or to any excipients of the study drug formulation.
15. Not able or willing to stop treatment with moderate or strong cytochrome P450 (CYP)3A4 inhibitors, or treatment with moderate or strong CYP3A4 inducers, within at least 1 week prior to Visit 3, until the end of treatment (the end of the run-out period).
16. Not able or willing to stop consumption of grapefruit, Seville (bitter) oranges or juices from those fruits within at least 1 week prior to Visit 3, and until the end of treatment (the end of placebo run-out period).
17. A prolonged QTc interval calculated using Fridericia's formula (QTcF) interval (QTcF greater than 450 ms). If the QTcF is greater than 450 ms on the first single 12-lead ECG, 2 additional 12-lead ECGs will be performed (at least after 30 min) and the mean of the 3 QTcF values will be calculated. (QTcF alculation formula seen in 11.5 Appendix)
18. Periodic limb movement disorder with arousal index (PLMAI)

    ≥ 15/h (assessed on the 1st PSG night), restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, or narcolepsy.
19. Apnea/hypopnea index ≥ 15/h according to American Academy of Sleep Medicine criteria or event associated with blood oxygen saturation level by pulse oximetry (SpO2) < 80%, as assessed on the 1st PSG night
20. A history of moderate to severe hepatic impairment (eg, Child-Pugh Class B or C). (details in 11.6 Appendix)
21. Sleep diary completed less than 70% between Visit 3 to Visit 4, or at least 3 days out of the 7 days immediately preceding the first PSG of visit 4.
22. Subjects who took placebo tablets less than 80% of days in from Visit 3 to Visit 4.

    Criteria assessed at Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5
23. Any of the following conditions related to suicidality:

    * Any suicidal ideation with intent, with or without a plan, at screening, i.e., answering "Yes" to questions 4 or 5 on the suicidal ideation section of the lifetime (Visit 1) and visit (Visit 2, Visit 3, Visit 4, Visit 5) version of the Columbia Suicide Severity Rating Scale© (C-SSRS©).
    * History of suicide attempt on the suicidal behavioral section of the lifetime version of the C-SSRS© (Visit 1).
24. Coronavirus Disease 2019 (COVID-19) positive subjects, supported by Antigen test or Nucleic acid detection.
25. For female subjects: pregnant, lactating or planning to become pregnant during projected duration of the study.
26. Positive urine drug test or presence of alcohol in exhaled breath as detected by breathalyzer test.
27. Unstable medical condition, significant medical disorder or acute illness, ECG, hematology or biochemistry test, thyroid function or coagulation test results within 1 month prior to the screening visit, which, in the opinion of the investigator, could affect the subject's safety or interfere with the study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline to month 1 in wake after sleep onset (WASO) measured by polysomnography(PSG). | Baseline to last 2 night(night 27 and 28)

SECONDARY OUTCOMES:
The change from baseline to the average of the last 7 days of month 1 in subjective total sleep time(sTST) measured by eDiary | Baseline to the average of the last 7 days of month 1
The change from baseline to month 1 in latency to persistent sleep (LPS) measured by PSG. | Baseline to last 2 night(night 27 and 28)

OTHER OUTCOMES:
Change from baseline to week 1 in the subjective total sleep time (sTST) measured by edairy. | Baseline to Week 1
Change from baseline to month 1 in the objective total sleep time (TST) measured by PSG. | Baseline to last 2 night(night 27 and 28)
Change from baseline to the last 7 days of month 1 in daytime functioning and alertness that is determined by scores on the visual analog scale (VAS ) at the end of the day. | Baseline to the average of the last 7 days of month 1
Change from baseline to Month 1 in wake after sleep onset (WASO) over time measured by PSG. | Baseline to last 2 night(night 27 and 28)
Change from baseline to the average of the last 7 nights of Month 1 in the subjective latency to sleep onset (sLSO) measured by eDiary. | Baseline to average of the last 7 days of Month 1
The change from baseline to week 1 in subjective latency to sleep onset (sLSO) measured by eDiary. | Base line to Week 1
Change from baseline to the last 7 nights of month 1 in subjective wake after sleep onset (sWASO) measured by eDiary. | Baseline to average of the last 7 days of month 1
The change from baseline to week 1 in subjective wake after sleep onset(sWASO) measured by eDiary. | Baseline to Week 1
Change from baseline to the last 7 days ofMonth 1/ Week 1 in sleep quality that is determined by scores on the visual analog scale(VAS) in the morning in eDiary. | Baseline to the average of the last 7 days of Month 1/ Week 1
Change from baseline to the last 7 days of Month 1/ Week 1 in depth of sleep that is determined by scores on the VAS (mm) in the morning in eDairy. | Baseline to the average of the last 7 days of Month 1/ Week 1
Change from baseline to the last 7 days of Month 1 / Week 1 in subjective number of awakenings measured by eDiary. | Baseline to the average of the last 7 days of Month 1/ Week 1
Change from baseline to Month 1 in Insomnia Severity Index (ISI) total score. ©) total score | Baseline to month 1
Change from baseline to Month 1 in sleep efficiency measured by PSG. | Baseline to month 1
The next-morning plasma concentrations 9-10 hours post dose at the first and second night of Visit 7 | Day 27/28 and Day 28/29

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Wang, Doctor, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (33):
- China (33):
  - The Second People's Hospital Of Hefei, Hefei, Anhui
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Chengdu Second People's Hospital, Chengdu, Chengdu
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Second Hospital of Suzhou University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - Deyang People's Hospital, Deyang, Sichuan
  - Tianjin Mental Health Center, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Seventh People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Wang H, Zhang B, Li C, Wang J, Xu L, Xu Q, Chen J, Xiao L, Wang Z, Wang B, Jiang Y, Liu Y, Yuan C, Ma Q, Wu J, Liu X, Huang Y, Cui H, Wang F, Wang Y. Efficacy and safety of daridorexant in Chinese patients with insomnia disorder: a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial. Sleep. 2025 Dec 11;48(12):zsaf170. doi: 10.1093/sleep/zsaf170. PMID 40557879